CLINICAL TRIAL: NCT00610298
Title: Effects of Whole Body Vibration in Elderly Patients Requiring Rehabilitation: A Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Another institution conducted and published this study.No subjects enrolled.
Sponsor: Ohio State University (Other)
Collaborators: Velimir Matkovic (Unknown)
Responsible Party: Principal Investigator, Lise Worthen-Chaudhari, Research Manager for Matkovic, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001H0215
Record Dates: First submitted 2007-12-26; First posted 2008-02-07 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Neuromuscular Deficits; Musculoskeletal Deficits
Keywords: disability affecting strength, balance and coordination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Subjects who receive whole body vibration
  Interventions: Device: whole body vibration using a Galileo vibrating platform
- N (No Intervention): Subjects do not receive whole body vibration intervention

INTERVENTIONS:
Device: whole body vibration using a Galileo vibrating platform — whole body vibration at 20 hertz for 3 minutes 3 to 5 days per week for up to 12 weeks
  Arms: I

SUMMARY:
The aim of this study is to accumulate data about the influence of whole body vibration on the functional recovery of adult patients with various neuromuscular and musculoskeletal deficits requiring physical medicine and rehabilitation treatments.

DETAILED DESCRIPTION:
We know that whole body vibration can cause remarkable increase in power in athletes, however, to what extent elderly and disabled individuals could benefit from it is currently unknown. Our primary goal is to investigate if treatment with whole body vibration in elderly persons and patients with various neuromuscular and musculoskeletal deficits would result in more rapid return of their function and presumably at a higher level than comparable group of patients undergoing standard physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* A history of one of the following conditions: CVA, Parkinson's disease, incomplete spinal cord injury, frail elderly, urinary incontinence, COPD, fibromyalgia
* Patients with neuromusculoskeletal problems affecting strength, balance, and coordination
* Must have all appendages (arms and legs) intact, not an amputee

Exclusion Criteria:

* Pregnancy
* Unable o participate in continuing outpatient therapy services at a location where the whole body vibration equipment is available
* Untreated deep venous thrombosis
* Other condition that will lead to poor treatment adherence
* History of join replacement of lower limbs, shoulders, or devices in the spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Berg Balance Test | begining and end of intervention

SECONDARY OUTCOMES:
Sit to stand test | begining and end of intervention
timed walking test | begining and end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Velimir Matkovic, M.D., Ph.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States